CLINICAL TRIAL: NCT07035015
Title: Self-Guided Immersive Virtual Reality Versus Mannequin-based Simulators to Teach the Ultrasound-Guided Supra-Inguinal Fascia Iliaca Block: A Non-inferiority Randomized Controlled Study
Brief Title: Self-Guided Immersive Virtual Reality Versus Mannequin-based Simulators to Teach the Ultrasound-Guided Supra-Inguinal Fascia Iliaca Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Yuqi Gu, Staff Anesthesiologist and Assistant Professor, The Ottawa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20240340-01H
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Nerve Block; Hip Fracture Surgeries
Keywords: Virtual Reality; Ultrasound-guided Regional Anesthesia; Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality UGRA (Experimental): The simulator applied principles of cognitive task analysis, which is a method aimed at describing the knowledge, cognitive process, and goal structures experts rely upon while performing a complex procedure
  Interventions: Other: VR UGRA
- Mannequin simulation (Active Comparator): The hybrid simulator will consist of a 3G mannequin and a gel-based part-task trainer.
  Interventions: Other: Mannequin-based simulation

INTERVENTIONS:
Other: VR UGRA — The simulator applied principles of cognitive task analysis, which is a method aimed at describing the knowledge, cognitive process, and goal structures experts rely upon while performing a complex procedure
  Arms: Virtual reality UGRA
Other: Mannequin-based simulation — The hybrid simulator will consist of a 3G mannequin and a gel-based part-task trainer.
  Arms: Mannequin simulation

SUMMARY:
This research project aims to see if using immersive virtual reality (iVR) is as good as using traditional mannequins to teach medical staff how to perform a specific nerve block called an ultrasound-guided supra-inguinal fascia iliaca (SIFI) block. This nerve block is important for managing pain in patients with hip fractures, as it can improve recovery, shorten hospital stays, and reduce healthcare costs. Currently, not enough eligible hip fracture patients receive these beneficial nerve blocks.

The study will recruit 36 staff and trainees from anesthesiology, emergency medicine, and orthopedic surgery at The Ottawa Hospital. Participants will be randomly assigned to one of two groups. One group will learn the SIFI block using a newly developed iVR simulator that uses real human anatomy and allows for practice of needling and injecting. The other group will use traditional mannequin-based simulators.

All participants will receive educational materials and videos before their training. Their skills will be tested before the training, immediately after, and again one month later using a hybrid simulator (a combination of a mannequin and a soft embalmed human cadaver part). The main thing being measured is their skill level using a standardized scoring system. The study also wants to see if the iVR simulator is well-tolerated by users. The overall goal is to improve care for hip fracture patients through better, more accessible training for medical staff.

DETAILED DESCRIPTION:
This research protocol outlines a single-center, non-inferiority randomized controlled trial (RCT) evaluating immersive virtual reality (iVR) against traditional mannequin-based, high-fidelity simulators (HFS) for training medical personnel in the ultrasound-guided supra-inguinal fascia iliaca (SIFI) block. This study addresses the suboptimal PNB utilization for hip fracture analgesia, despite evidence supporting their benefits, with fewer than 20% of eligible patients in Ontario and at The Ottawa Hospital (TOH) receiving them due to institutional or provider factors.

The primary scientific objective is to ascertain if the novel iVR UGRA simulator, featuring veridical human anatomy and real-time simulated interaction, is non-inferior to HFS for imparting SIFI block skills. Secondary endpoints include assessing iVR tolerability (cybersickness, cognitive load) and collecting formative data for platform iteration.

The study cohort will be 36 (target N=40) TOH medical staff and trainees (anesthesiology, emergency medicine, orthopedics), excluding those with >5 SIFI blocks/year or advanced regional anesthesia training. After informed consent and baseline DASS-21 collection, participants undergo stratified randomization (specialty, PGY level) to the VRS or HFS arm.

Both groups receive standardized didactics (SIFI text, videos on ultrasound, needling, sonoanatomy) followed by 60 minutes of self-directed practice with a checklist. The HFS group uses a 3G mannequin and gel part-task trainer. The VRS group uses the VitaSim iVR simulator (designed with cognitive task analysis and functional task alignment), which currently lacks tactile feedback and patient communication modules.

Skill assessment occurs pre-intervention, immediately post-intervention, and at a 1-month retention interval, involving SIFI block performance on a hybrid simulator (mannequin/Thiel cadaveric model). Performances are video-recorded for blinded, independent rating by two calibrated assessors. The primary outcome is the UGRA Global Rating Scale (GRS) score. Secondary outcomes include checklist scores, procedural duration, needle passes, simulated IM injections, practice time, and for the VRS group, scores on presence, cognitive load, and cybersickness questionnaires.

Sample size (12 per discipline) is based on a non-inferiority margin of 7.6 on the GRS (α=0.05, power=0.9). Statistical analyses via SPSS will include descriptive/inferential statistics (Shapiro-Wilk, t-tests/Wilcoxon, ANCOVA for primary outcome controlling for baseline GRS). Inter-rater reliability uses intraclass correlation coefficients (ICC); significance is p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Staff and trainees from anesthesiology, emergency medicine, and orthopedic surgery. All participants will be locally recruited within The Ottawa Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Guided Regional Anesthesia Global Rating Scale | From enrolment until the 1 month retention.
  The primary outcome is the summation of the UGRA Global Rating Scale (GRS), which is a valid assessment tool to score trainees' performance in UGRA. Previous studies have found a strong correlation in the GRS score between simulated and real clinical settings. The minimum score is 9 and maximum score is 35. A high score represents better procedural performance.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No